CLINICAL TRIAL: NCT00917163
Title: A Randomized Comparison of the Supralimus® Stent With the Xience V™ Stent in the Treatment of Patients With de Novo Native Coronary Artery Lesions
Brief Title: SERIES III RUN-IN Clinical Trial: A Comparison of the Supralimus® Stent With the Xience V™ Stent
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: due to unavoidable circumstances relating to logistic issues and regulatory processes in various countries causing unacceptable delays.
Sponsor: Sahajanand Medical Technologies Limited (Industry)
Collaborators: Cardialysis BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SES/RCT/01
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; restenosis; stent thrombosis; coronary stents; angioplasty; drug eluting stents
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supralimus(R) Sirolimus Eluting Stent (Experimental): Supralimus® Coronary Stent System consisting of the MATRIX® Coronary Stent having Sirolimus eluting from Biodegradable Polymeric Matrix on a Stainless Steel Platform, Drug concentration 1.4 µg/mm2
  Interventions: Device: Supralimus(R) Sirolimus-Eluting Coronary Stent System
- Xience V™ Everolimus Eluting Stent (Active Comparator): The XIENCE V™ Everolimus Eluting Coronary Stent System consisting of the MULTI-LINK VISION® Coronary Stent System coated with a formulation containing everolimus, the active ingredient, embedded in a non-erodible polymer., Drug Load: 100 µg/cm2
  Interventions: Device: Xience V™ Everolimus Eluting Coronary Stent

INTERVENTIONS:
Device: Supralimus(R) Sirolimus-Eluting Coronary Stent System — Drug eluting stent implantation in the treatment of coronary artery disease.
  Other Names: Drug Eluting Stent
  Arms: Supralimus(R) Sirolimus Eluting Stent
Device: Xience V™ Everolimus Eluting Coronary Stent — Drug eluting stent implantation in the treatment of coronary artery disease
  Other Names: Drug Eluting Stent
  Arms: Xience V™ Everolimus Eluting Stent

SUMMARY:
The objective of Series III Run-In Trial is to compare the performance and efficacy of the Supralimus® sirolimus-eluting stent with the Xience V™ everolimus-eluting stent with respect to in-stent luminal late loss at 9 months as assessed by off-line QCA. Ninety percent power to reject the null hypothesis that the Supralimus® stent is inferior to Xience V™ in favor of the alternative hypothesis that the Supralimus® stent is not inferior to Xience V™.

DETAILED DESCRIPTION:
Series III Run-In is a prospective, multi-center, randomized, single-blind (patient-blind), non-inferiority trial to be conducted at approx. 35 interventional cardiology centers in India, Brazil, Argentina, Thailand and Saudi Aurabia. A total of 360 will be randomized on a 2:1 basis to either the Supralimus® (sirolimus-eluting) stent or the Xience V™ (everolimus-eluting) stent.

In selected sites, IVUS will also be recorded in these patients (maximum of 60 IVUS patients in total), at baseline (post-procedure) and at 9-month follow-up.

All patients will be followed clinically for up to 5 years after stent implantation. Repeat angiography will be performed in all patients at 9 months after the index procedure.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥18 years.
2. Eligible for percutaneous coronary intervention (PCI)
3. Acceptable candidate for CABG
4. Clinical evidence of ischemic heart disease and/or a positive territorial functional study. Documented stable angina pectoris ((Canadian Cardiovascular Society (CCS) Classification 1, 2, 3 or 4) or unstable angina pectoris with documented ischemia (Braunwald Class IB-C, IIB-C or IIIB-C), or documented silent ischemia.
5. The target lesion is a single de novo coronary artery lesion with ≥ 50% and < 100% stenosis in one of the major epicardial territories (LAD, LCX or RCA). A second target lesion in another major epicardial vessel could be treated and this second lesion should fit with the inclusion/exclusion criteria and will receive the same type of stent.
6. The target lesion must be covered by one study stent, preferably with a margin of 3 mm on each side of the lesion.
7. The target lesion must be ≤ 22 mm in length by visual estimate.
8. The target reference vessel diameter must be ≥ 2.5 mm and ≤ 3.5 mm.
9. Patient or patient's legal representative has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee of the clinical site.

Exclusion Criteria:

1. Female of childbearing potential
2. Documented left ventricular ejection fraction (LVEF) ≤ 30%
3. Evidence of an acute Q-wave or non-Q-wave myocardial infarction within 72 hours preceding the index procedure
4. Known allergies to the following: aspirin, clopidogrel bisulfate (Plavix®, Ceruvin) or ticlopidine (Ticlid®), heparin, sirolimus, everolimus, stainless steel, cobalt, chromium, contrast agent (that cannot be adequately pre-medicated)
5. A platelet count <100,000 cells/mm3 or >700,000 cells/mm3 or a WBC <3,000 cells/mm3
6. Acute or chronic renal dysfunction (creatinine >2.0mg/dl or >150µmol/L)
7. Total occlusion (TIMI 0) or TIMI 1
8. Target vessel has evidence of thrombus
9. Target vessel is excessively tortuous which makes it unsuitable for proper stent delivery and deployment
10. Previous bare metal stenting (less than 1 year) anywhere within the target vessel
11. Previous drug-eluting stenting anywhere within any epicardial vessel
12. The target lesion requires treatment with a device other than PTCA prior to stent placement (e.g. but not limited to, directional coronary atherectomy, excimer laser, rotational atherectomy, etc.)
13. Significant (>50%) stenosis proximal or distal to the target lesion that might require revascularization or impede run-off
14. Heavily calcified lesion and/or calcified lesion which cannot be successfully predilated
15. Target lesion is located in or supplied by an arterial or venous bypass graft
16. Ostial target lesion
17. Target lesion involves a side branch >2.0mm in diameter with an ostial disease
18. Patient is currently participating in an investigational drug or device study, including its follow-up period
19. Within 30 days prior to procedure, patient has undergone a previous coronary interventional procedure of any kind
20. Within 60 days post-procedure, patient requires planned interventional treatment of any non-target vessel. Planned intervention of the target vessel after the index procedure is not allowed.
21. Stroke or transient ischemic attack within the prior 6 months
22. Unprotected Left Main (LM) coronary artery disease (stenosis >50%)
23. In the investigator's opinion, patient has a co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study
24. Planned surgery within 6 months after the index procedure
25. Life expectancy less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
In-stent luminal late loss at 9 months after stent implantation (off-line QCA). | 9 months

SECONDARY OUTCOMES:
PROCEDURAL: Pre-procedure Syntax Score (by off-line visual assessment), Procedural success rate, Device success rate | Hospital discharge
ANGIOGRAPHIC : Minimal lumen diameter (MLD), % diameter stenosis, In-segment late loss, Proximal late loss, Distal late loss, Binary restenosis rate | 9 months
IVUS (in a subset of patients): Minimal lumen area, Vessel volume, Lumen volume, Neointimal hyperplasia, Volume obstruction, Incomplete stent apposition, Plaque behind the stent struts | 9 months
DEVICE-ORIENTED COMPOSITE ENDPOINT : Cardiac death, MI not clearly attributable to a non-target vessel, Target lesion revascularization (TLR) | 30 days, 6 months, 9 months, 1, 2, 3, 4, and 5 years
PATIENT-ORIENTED COMPOSITE ENDPOINT : All-cause death, Any MI (including non-target vessel territory), Any repeat revascularization (including all target and non-target vessel) | 30 days, 6 months, 9 months, 1, 2, 3, 4, and 5 years
STENT THROMBOSIS | 30 days, 6 months, 9 months, 1, 2, 3, 4, and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Patrick W Serruys, MD, Ph.D, Study Chair — Thoraxcenter,Rotterdam,NL
Locations (28):
- Brazil (13):
  - Incor Hospital, Brasília, Brasília
  - Hospital Meridional, Vitaria, Espírito Santo
  - Centro de Cardiologia e Radiologia Intervencionista, Goiânia, Goiás
  - Cardiovascular Diagnóstico, Campo Grande, Mato Grosso do Sul
  - Santa Casa de misericórdia de Juiz de fora, Juiz de Fora, Minas Gerais
  - Intistuto do Coracao do Triangulo, Uberlândia, Minas Gerais
  - Hospital Costantino Constantini, Curitiba, Paraná
  - Instituto de Cardiologia, São Paulo, São Paulo
  - Hospital Bandeirantes, São Paulo, São Paulo
  - Incor Hospital, São Paulo, São Paulo
  - Instituto Dante Pazzanese, São Paulo, São Paulo
  - Hospital Albert Einstein, São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo, São Paulo
- India (14):
  - Life Care Institute, Ahmedabad, Gujarat
  - Shri.Jayadeva Institute of Cardiology, Bangalore, Karnataka
  - P.R.S Hospital, Trivandrum, Kerala
  - Jaslok Hospital & Research Centre, Mumbai, Maharashtra
  - KEM Hospital, Mumbai, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Escorts Heart Institute & Research Centre, New Delhi, National Capital Territory of Delhi
  - Max Devki Devi Heart and Vascular Institute, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Apollo Hospital, Chennai, Tamil Nadu
  - Madras Medical Mission, Chennai, Tamil Nadu
  - Sanjay Gandhi Post Graduate Institute of Medical Sciences, Lucknow, Uttar Pradesh
  - Kailash Health Care Limited, Noida, Uttar Pradesh
  - B.M.Birla Heart Research Center, Kolkata, West Bengal
- KAUH King Abdl Aziz University Hospital, Jeddah, Saudi Arabia

REFERENCES:
- [Background] Dani S, Kukreja N, Parikh P, Joshi H, Prajapati J, Jain S, Thanvi S, Shah B, Dutta JP. Biodegradable-polymer-based, sirolimus-eluting Supralimus stent: 6-month angiographic and 30-month clinical follow-up results from the series I prospective study. EuroIntervention. 2008 May;4(1):59-63. doi: 10.4244/eijv4i1a11. PMID 19112780
- [Background] Dr. A.Abhyankar; Evaluation of Safety, Efficacy and Procedural Outcomes of Extra Long Sirolimus Eluting Stent with novel polymeric technology for treatment of long de novo coronary lesions; Catheterization Cardiovascular Interventions; 3rd Nov - 2nd Dec 2006; DOI 10.1002/ccd.21033